CLINICAL TRIAL: NCT01307943
Title: Mindfulness-based Stress Reduction for Pediatric Mental Health
Acronym: MBSR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: CASA: Child, Adolescent and Family Mental Health (Unknown)
Responsible Party: Principal Investigator, Sunita Vohra, Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBSR1
Record Dates: First submitted 2011-02-25; First posted 2011-03-03 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Mental Health Wellness 1
Keywords: MBSR; adolescent; mental health
MeSH Terms: conditions — Psychological Well-Being | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness Based Stress Reduction (Experimental): Eight MBSR sessions of 2 hrs/week to be held during regular class time plus one 3-hour retreat at the completion of the eight sessions to review and consolidate experience with the various mindfulness practices. The MBSR concepts and techniques will emphasize portability. Participants will be encouraged to find moments throughout their day in which to practice the techniques. The language used to describe mindfulness practices will be accessible to youth. Mindfulness concepts will be linked with tag phrases like "breathing break," "autopilot," and "choice points." Homework will emphasize experiential, concrete tasks ("notice five new things today"; "eat one meal mindfully this week").
  Interventions: Other: Mindfulness-based stress reduction program
- Usual Care (Active Comparator): The control group will be youth receiving therapies and programs already used at the site. The site provides family centered treatment where adolescents take part in therapy from Sunday evening until Friday afternoon. In addition to a structured day and evening schedule, standard treatment includes: Daily group therapy; ii) Medications; iii) Schooling by Edmonton Public School Board teachers; iv) Physical education and recreation; and v) Weekly Multiple Family Therapy.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Mindfulness-based stress reduction program — Eight MBSR sessions of 2 hrs/week to be held during regular class time plus one 3-hour retreat
  Other Names: MBSR
  Arms: Mindfulness Based Stress Reduction
Other: Usual care — The site provides family centered treatment where adolescents take part in therapy from Sunday evening until Friday afternoon. In addition to a structured day and evening schedule, standard treatment includes: Daily group therapy; ii) Medications; iii) Schooling by Edmonton Public School Board teachers; iv) Physical education and recreation; and v) Weekly Multiple Family Therapy.
  Other Names: standard care
  Arms: Usual Care

SUMMARY:
Mindfulness-based stress reduction (MBSR) is a group program in which participants are taught to be mindful or present-focused. MBSR programs consist of instruction in a variety of mindfulness meditations including body scan, sitting meditation, mindful yoga, and discussion of these practices. Our study purpose is to develop and conduct a pilot mixed-methods randomized controlled trial (RCT), combining clinical outcomes, qualitative interviews, and brain imaging to assess the impact of the intervention on children with mental health challenges.

DETAILED DESCRIPTION:
This study will be a 2 arm controlled clinical trial (CCT) comparing usual care to usual care plus MBSR. Participants will be residents of a local inpatient treatment facility for adolescents with serious mental health issues. Outcomes the investigators will measure include mental health status as well as mindfulness. The investigators will also conduct qualitative interviews to assess the personal impact of the intervention on the patients and their families. In order to map and measure cognitive changes during MBSR the investigators will conduct brain imaging using functional magnetic resonance imaging (fMRI) and Event-Related Potential (ERP) recordings. Through this study the investigators will determine if MBSR is helpful to our population.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 12 and 18
* residents of study site
* communication and comprehension of English
* not currently abusing substances

Exclusion Criteria:

* participants diagnosed with psychosis, as meditation has rarely been associated with precipitation of psychosis and/or psychotic episodes in individuals with pre-existing schizophrenia or significant thought disorders

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Behavioral Assessment System for Children - 2nd Edition | change from baseline at 10 weeks after start of intervention (or control period)

SECONDARY OUTCOMES:
Child Acceptance and Mindfulness Measure (CAMM) | change from baseline at 10 weeks after start of intervention (or control period)
EEG and fMRI | change from baseline at 10 weeks after start of intervention (or control period)
Adverse events | at any stage during the study
Qualitative interview | 12 weeks after start of intervention
  this will occur only for intervention group
Emotion regulation in childhood and adolescence(ERQ-CA) | change from baseline at 10 weeks after start of intervention (or control period)
Behavioral Assessment System for Children - 2nd Edition | change from baseline 3 months after intervention is complete and same time frame for control group
Child Acceptance and Mindfulness Measure (CAMM) | change from baseline 3 months after intervention is complete and same time frame for control group
Emotion regulation in childhood and adolescence(ERQ-CA) | change from baseline 3 months after intervention is complete and same time frame for control group
Perceived Stress Scale (PSS) | change from baseline at 10 weeks after start of intervention (or control period)
Perceived Stress Scale (PSS) | change from baseline 3 months after intervention is complete and same time frame for control group

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Vohra, MD, MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Vohra S, Punja S, Sibinga E, Baydala L, Wikman E, Singhal A, Dolcos F, Van Vliet KJ. Mindfulness-based stress reduction for mental health in youth: a cluster randomized controlled trial. Child Adolesc Ment Health. 2019 Feb;24(1):29-35. doi: 10.1111/camh.12302. Epub 2018 Oct 15. PMID 32677243